CLINICAL TRIAL: NCT06767176
Title: Impact of Dietary Nitrate Supplementation on VO2max During Ramadan Fasting in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Philip Millar, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25-01-006
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Ramadan Fasting
Keywords: Ramadan; Fasting; VO2max; Dietary Nitrate
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): Normal Fasting, no intervention. During this arm, participants will be asked to complete an exercise test before and after 1 week of Ramadan fasting.
- Nitrate Supplementation (Experimental): Participants will be asked to consume daily nitrate supplementation (70ml) in the form of beetroot juice for 7 days. Participants will then complete a maximal exercise test as they fast.
  Interventions: Dietary Supplement: Beetroot Juice (Beet-It Stamina Shot) & Supervised Exercise Training

INTERVENTIONS:
Dietary Supplement: Beetroot Juice (Beet-It Stamina Shot) & Supervised Exercise Training — 7 doses, taken daily, 70 ml shots, consumed in the morning before the start of fasting
  Arms: Nitrate Supplementation

SUMMARY:
The goal of this clinical trial is to determine if beetroot juice supplementation changes exercise performance following one week of Ramadan fasting in young, healthy adults. The main question it aims to answer is:

Does daily beetroot juice supplementation change VO2 max in fasting individuals during the first week of Ramadan?

Participants will:

Visit the lab before the start of Ramadan and after one week of fasting If assigned to intervention group, consume daily shots of beetroot juice (70ml) during the first week of Ramadan fasting Perform maximal exercise testing on a cycle ergometer

DETAILED DESCRIPTION:
Recent literature demonstrates data showing a decrease in VO2max during the first week of Ramadan fasting. This is a practice observed by millions around the world every year, where individuals abstain from food and water from sunrise to sunset, dictated by the lunar calendar. Dietary nitrate consumption has been shown to increase VO2max and exercise performance. Therefore, the primary purpose of this study is to investigate whether dietary nitrate, in the form of beetroot juice, can help mitigate the decrease in VO2 max during the first week of Ramadan fasting.

24 young healthy adults will be recruited to undergo these two visits. The first visit will assess maximal oxygen uptake to determine aerobic fitness and metabolic exercise intensity zones under non-fasting conditions. The second visit will be completed after one week of Ramadan fasting. If assigned to the intervention group, participants will consume one shot (70ml) of Blonyx - Beet It Sport Nitrate 400 beetroot juice every day. Each shot contains 400mg of nitrates. Urine Specific Gravity will be measured after each visit to assess hydration status. The intervention group will also undergo Single Blood Draws after each visit to assess nitrate concentrations before and after a week of consumption.

ELIGIBILITY:
Inclusion Criteria:

* Free of known cardiovascular or metabolic diseases or sleep disorders
* No history of smoking (within the past 3 months)
* Able to engage in physical activity assessed through the physical activity readiness questionnaire (PAR-Q+)
* No prescription of chronic medications other than oral contraceptives
* Able to abide by fasting protocols for all visits
* Individuals who are not allergic to ultrasound gel or beetroot juice
* Individuals who are not pregnant

Exclusion Criteria:

* Individuals diagnosed with cardiovascular or metabolic disease or sleep disorders
* Has a history of smoking (within the past 3 months)
* Not ready to engage in physical activity as assessed by the PAR-Q+
* Individuals prescribed chronic medications other than oral contraceptives
* Unable to abide by fasting protocols for any testing visit
* Allergic to ultrasound gel or beetroot juice
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
VO2 max | One--week differences between before and after 1 week of fasting, nitrate supplementation if in intervention group
  Maximal Oxygen Uptakes will be assessed to analyze aerobic capacity and fitness under fasting conditions.

SECONDARY OUTCOMES:
Nitrate Concentration levels | Comparison between blood before and after nitrate supplementation: one week
  Single blood draws will be taken after each visit for the nitrate supplementation group

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Millar, PhD, Principal Investigator — University of Guelph

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Time Frame: Beginning after publication with no end date
Access Criteria: Phillip Millar, University of Guelph

REFERENCES:
- See also: Intervention Wesbite. — https://blonyx.ca/pages/subscribe-save